CLINICAL TRIAL: NCT05177523
Title: INsIDER: Imaging the Interplay Between Axonal Damage and Repair in Multiple Sclerosis
Brief Title: Imaging the Interplay Between Axonal Damage and Repair in Multiple Sclerosis
Acronym: INsIDER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01174; me18Granziera
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis (MS); Relapsing-remitting Multiple Sclerosis (RRMS); Secondary-progressive Multiple Sclerosis (SPMS); Primary Progressive Multiple Sclerosis (PPMS)
Keywords: axonal damage; axonal demyelination; axonal degeneration; axonal loss; axonal disorganization; axonal repair; axonal remyelination; axonal reorganization; Advanced MRI (aMRI); Neurite Orientation Dispersion and Density Imaging (NODDI); Diffusion Kurtosis (DK); Magnetization Transfer Imaging (MTI); Multi-echo Susceptibility-Based imaging (SBI); Myelin Water Imaging (MWI); T1 relaxometry (quantitative T1, qT1); machine learning technique
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be coded at acquisition and then aliquoted and stored at - 75 C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS patient group: Recruitment of 200 MS patients at the MS Clinic of the Department of Neurology (Neurologische Klinik und Poliklinik), University Hospital Basel (Universitätsspital Basel)
  Interventions: Diagnostic Test: MRI; Other: blood sampling
- control group (HC): Recruitment of 100 healthy controls (HC) by public announcements (i.e. advertisement/flyer) on the University Hospital's and the University's notice board.
  Interventions: Diagnostic Test: MRI; Other: Neurocognitive examination for healthy subjects; Other: blood sampling

INTERVENTIONS:
Diagnostic Test: MRI — Each enrolled subject will undergo a MRI at baseline and a second MRI at 2 years (+/- 3 months) follow-up.
Other: Neurocognitive examination for healthy subjects — Neurocognitive examination for healthy subjects will be performed at both baseline and follow-up
  Groups: control group (HC)
Other: blood sampling — Each enrolled subject will undergo a blood sampling (10 ml) at baseline

SUMMARY:
This project is to:

1. Quantify differences in axonal integrity and organization in aMS versus naPMS patients.
2. Quantify changes in axonal integrity and organization in aMS versus naPMS patients over a two-year period.
3. Validate the combination of imaging parameters that best differentiate aMS versus naPMS patients using histopathology.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system characterized by multifocal inflammatory infiltrates, microglial activation and degradation of oligodendrocytes, myelin and axons. Clinical MS categories exhibit variable amount of central nervous system (CNS) damage and repair, depending on numerous variables including genetic, immunological, pathological and environmental factors.

Therefore, understanding the interplay between axonal damage (i.e. axonal demyelination/degeneration/loss/disorganization) and (ii) axonal repair (i.e. axonal remyelination/reorganization) in living MS patients may be the key to understand disease progression, to establish accurate disease monitoring criteria and to predict disease response to future reparative therapies. New in-vivo methods are necessary to elucidate the interplay between axonal damage and repair in the brain of living patients with MS. Advanced MRI (aMRI) permits a multifaced quantification of the various components of the axons and their organization. Neurite Orientation Dispersion and Density Imaging (NODDI) and Diffusion Kurtosis (DK) are new approaches in clinical research This study is to identify in vivo the specific neuropathological pattern of axonal damage and repair exhibited by active MS (aMS) and non-active progressive MS (naPMS) patient by leveraging the information provided by model-based diffusion metrics (NODDI, DK), Magnetization Transfer Imaging (MTI), Multi-echo Susceptibility-Based imaging (SBI), Myelin Water Imaging (MWI) and quantitative T1 relaxometry (qT1). These advanced MRI contrasts provide complementary and partially redundant information about the axonal structure and its organization (i.e. density and orientation of axons and dendrites in the brain tissue, axonal integrity and myelination, presence of myelin and iron, and brain tissue architecture). Therefore, their combination may prove high sensitivity and specificity to axonal damage and repair.

This project has 3 main aims:

Aim 1. Quantify differences in axonal integrity and organization in aMS versus naPMS patients.

Aim 2. Quantify changes in axonal integrity and organization in aMS versus naPMS patients over a two-year period.

Aim 3. Validate the combination of imaging parameters that best differentiate aMS versus naPMS patients using histopathology.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patients may be diagnosed with:

  1. active RRMS (n=100): Relapsing-remitting course and > 1 clinical relapse and/or signs of MRI activity (> 1 Gd enhancing lesion) during the last year before study enrollment.
  2. non-active PMS (n=100): Progressive course (PPMS or SPMS) and no clinical relapses and/or signs of MRI activity during the last year before study enrollment.
* Age 18-80 years old
* No other neurological or psychiatric disorder

Inclusion criteria for healthy controls:

* Age 18-80 years old
* No other neurological or psychiatric disorder

Exclusion Criteria for patients and healthy controls:

* Pregnancy
* Contraindication to MRI (eg, claustrophobia, metallic implants, pacemaker etc).
* Inability to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruitment of MS patients will take place at the MS Clinic of the Department of Neurology (Neurologische Klinik und Poliklinik), University Hospital Basel (Universitätsspital Basel). Healthy subjects will be recruited by public announcements (i.e. advertisement/flyer) on the University Hospital's and the University's notice board.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
MRI- change in axonal integrity and organization over 2 years in aMS, naPMS and HC, by using machine learning techniques | at baseline and 2 years (+/- 3 months) after baseline
  After magnetic resonance (MR) data preprocessing (image denoising, standardization, bias field correction) classical machine learning techniques will be used to classify a number of MRI metrics which will be averaged over a number of regions of interest (ROIs) including (i) normal-appearing white and brain matter in brain lobes and cervical spinal cord, (ii) basal ganglia, (iii) thalamus, (vi) cerebellum, MS lesions. Complex input data (voxels/patches) will be generated to learn from, then a deep learning model for supervised classification will be defined to identify the combination of aMRI parameters that characterize aMS, naPMS and HC.

SECONDARY OUTCOMES:
Change in MUSIC Test | at baseline and 2 years (+/- 3 months) after baseline
  Neurocognitive examination. MUSIC is a rapid (about 10-12 min) multiple domain cognitive screening test reflecting the most frequently impaired cognitive domains in MS. At 20-30 points the performance is in the normal range, at 16-19 points there is at most slight cognitive dysfunction, at 11-15 points there is moderate cognitive dysfunction and at <= 10 points there is a clear cognitive dysfunction.
Change in auditory verbal learning and memory test/ Verbaler Lern- und Merkfähigkeitstest (VLMT) | at baseline and 2 years (+/- 3 months) after baseline
  Questionnaire to investigate memory performance, learning and recall information. Five presentations of a 15-word list are given, each followed by attempted recall. This is followed by a second 15-word interference list (list B), followed by recall of list A. Delayed recall and recognition are also tested.
Change in Symbol Digital Modalities Test (SDMT) | at baseline and 2 years (+/- 3 months) after baseline
  The SDMT detects cognitive impairment by measuring the time to pair abstracts. Using a reference key, the test taker has 90 seconds to pair specific numbers with given geometric figures.
Change in Brief Visuospatial Memory Test (BVMT) | at baseline and 2 years (+/- 3 months) after baseline
  The BVMT measures visuospatial memory In three Learning Trials, the respondent views the stimulus page for 10 seconds and is asked to draw as many of the figures as possible in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Last, a Recognition Trial, in which the respondent is asked to identify which of 12 figures were included among the original geometric figures, is administered. Slower processing speed is associated with poorer learning and memory performance.
Change in Hospital Anxiety and Depression Scale (HADS) | at baseline and 2 years (+/- 3 months) after baseline
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Granziera, Prof. Dr. med., Principal Investigator — Department of Neurology, University Hospital Basel
Locations (1):
- University Hospital Basel, Department of Neurology, Basel, Switzerland